CLINICAL TRIAL: NCT06310876
Title: A Phase 1 Placebo-and Active-Controlled Crossover Study of the Potential for Cardiac Repolarization Effects Following Single Dose of ABBV-CLS-7262 in Healthy Subjects
Brief Title: A Thorough QT Study of ABBV-CLS-7262 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calico Life Sciences LLC (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: M24-852
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: TQT; Pharmacokinetics
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Subjects will receive ABBV-CLS-7262 dose 1, ABBV-CLS-7262 dose 2, placebo, or moxifloxacin 400 mg tablet
  Interventions: Drug: ABBV-CLS-7262; Drug: Placebo; Drug: Moxifloxacin 400mg
- Sequence 2 (Experimental): Subjects will receive ABBV-CLS-7262 dose 1, ABBV-CLS-7262 dose 2, placebo, or moxifloxacin 400 mg tablet
  Interventions: Drug: ABBV-CLS-7262; Drug: Placebo; Drug: Moxifloxacin 400mg
- Sequence 3 (Experimental): Subjects will receive ABBV-CLS-7262 dose 1, ABBV-CLS-7262 dose 2, placebo, or moxifloxacin 400 mg tablet
  Interventions: Drug: ABBV-CLS-7262; Drug: Placebo; Drug: Moxifloxacin 400mg
- Sequence 4 (Experimental): Subjects will receive ABBV-CLS-7262 dose 1, ABBV-CLS-7262 dose 2, placebo, or moxifloxacin 400 mg tablet
  Interventions: Drug: ABBV-CLS-7262; Drug: Placebo; Drug: Moxifloxacin 400mg

INTERVENTIONS:
Drug: ABBV-CLS-7262 — • single oral Dose 1
Drug: ABBV-CLS-7262 — • single oral Dose 2
Drug: Placebo — • single oral dose
Drug: Moxifloxacin 400mg — • single oral dose

SUMMARY:
This is a randomized, blinded, placebo and active-controlled, 4-period, crossover design thorough QT/QTc (TQT) study to evaluate the effect of ABBV-CLS-7262 on cardiac repolarization in healthy adult subjects.

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo and active-controlled, 4-period, crossover study. The study will be double-blinded for ABBV-CLS-7262 (dose 1 or dose 2) and placebo regimens and open-label for moxifloxacin. 72 subjects are planned to be enrolled.

All subjects will receive a single oral dose of 4 different study treatments over 4 separate treatment periods, each separated by a washout period.

On Day 1 of each period, subjects will receive either ABBV-CLS-7262 dose 1, ABBV-CLS-7262 dose 2, placebo, or moxifloxacin 400 mg.

In each period, cardiodynamic ECGs will be collected pre-dose and for 24 hours post-dose and PK blood samples will be collected pre-dose and for 48 hours post-dose. Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers in general good health.
* Must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.
* Individuals between 18 and 55 years of age inclusive at the time of screening.
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 29.9 kg/m2
* All male subjects who are sexually active and not surgically sterilized must agree to use an acceptable contraceptive method. Additionally, male subjects must agree to not donate sperm during the study until 30 days after the final dose of study drug.
* All female subjects who are sexually active and of childbearing potential must agree to use a highly effective contraceptive method. Additionally, female subjects must agree to not donate eggs during the study and for 30 days after the final dose of study drug.

Exclusion Criteria:

* Subject who, in the opinion of the investigator, is incapable of completing study-required visits and procedures
* Pregnant or breastfeeding.
* Treatment with any other investigational treatment within 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of ABBV-CLS-7262 on the QTc interval in healthy adult subjects | Up to 24 hours
  To evaluate the effect of ABBV-CLS-7262 on the QTc interval in healthy adult subjects.

SECONDARY OUTCOMES:
To evaluate the effects of ABBV-CLS-7262 on change in electrocardiogram (ECG) parameters | Up to 24 hours
  ECG parameters include RR and PR interval, QRS duration and heart rate (HR).
To evaluate the sensitivity of QTc measurement using moxifloxacin | Up to 24 hours
  To evaluate the sensitivity of QTc measurement using moxifloxacin.
To evaluate the effect of ABBV-CLS-7262 on T-wave morphology | Up to 24 hours
  To evaluate the effect of ABBV-CLS-7262 on T-wave morphology.

CONTACTS AND LOCATIONS:
Locations (1):
- AbbVie Clinical Pharmacology Research Unit (ACPRU), Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No